CLINICAL TRIAL: NCT00900510
Title: The Use of Adjuvant Antibiotic Therapy After Incision and Drainage for Pediatric Abscess: A Prospective, Randomized, Double-blinded, Placebo-Controlled Trial
Brief Title: Antibiotic Therapy After Incision and Drainage for Abscess
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment of this population in the hospital setting not practical.
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00008450
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2014-12

CONDITIONS: Abscess
Keywords: subcutaneous abscess; Incision and drainage; Methicillin-resistant staphylococcus aureus
MeSH Terms: conditions — Abscess; Surgical Wound | interventions — Drainage; Trimethoprim; Sulfamethoxazole; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drainage and placebo (Experimental): Incision and drainage with placebo.
  Interventions: Procedure: Incision and drainage; Drug: Placebo
- Drainage with TMP/SX (Active Comparator): Drainage with Bactrim
  Interventions: Drug: Trimethoprim/Sulfamethoxazole (Bactrim)

INTERVENTIONS:
Procedure: Incision and drainage
  Arms: Drainage and placebo
Drug: Trimethoprim/Sulfamethoxazole (Bactrim) — Trimethoprim/Sulfamethoxazole, oral
  Arms: Drainage with TMP/SX
Drug: Placebo
  Arms: Drainage and placebo

SUMMARY:
Background: Skin abscesses are a growing problem in the general pediatric population around the world. While the standard treatment for an abscess/boil is incision and drainage, many physicians also prescribe antibiotics, despite the lack of evidence that antibiotics are necessary to help the wound heal. The purpose of this research study is to determine whether antibiotics are necessary after incision and drainage of a skin abscess in children. This is an important question because medical evidence has shown that using antibiotics when they are not needed has contributed to the increase of bacterial antibiotic resistance. In fact, several of the antibiotics that successfully killed Staph bacteria several years ago are now no longer effective because of antibiotic resistance. Now resistant forms of Staph bacteria, called "Community-Acquired Methicillin-Resistant Staph Aureus" (CA-MRSA), account for 50-85% of all pediatric skin abscesses. If antibiotics are not necessary then withholding them when appropriate may help slow the progression of antibiotic-resistant Staph infections.

Objective(s) and Hypothesis(es): The investigators believe that antibiotics are no better than placebo at achieving a cure after drainage of an abscess in a child. The objective of this study is to answer the question: Do antibiotics after abscess drainage result in a better chance of cure than placebo?

Potential Impact: If abscess drainage alone is shown to be as effective as drainage followed by antibiotics, then the routine use of antibiotics for this problem could be avoided. This would help limit the increasing antibiotic resistance of bacteria (especially CA-MRSA) in communities around the world. A well-designed study may provide the evidence to change the way children are treated for abscesses in a future where antibiotic resistant bacteria will be even more of a public health challenge.

ELIGIBILITY:
Inclusion Criteria:

* Any child (age 6 months-18 years old) that:

  * does not meet criteria for hospitalization and
  * has only one localized abscess (>/= 2 cm of erythema and induration), which is clinically judged to be amenable to incision and drainage. (i.e., on clinical exam their is fluctuance, erythema, induration, and/or purulent drainage)
  * has an abscess that is ± 7 days from onset, who requires surgical incision and drainage for a skin and soft-tissue abscess

Exclusion Criteria:

* children < 6 months of age
* children who require inpatient hospitalization - children with a medical condition in which adjuvant antibiotic therapy would be accepted standard of practice (i.e., history of neutropenia, cardiac surgery, indwelling prosthesis)
* children with a previously diagnosed immunodeficiency (HIV, Chronic Granulomatous Disease, Job's syndrome, chronic steroid use)
* children hospitalized within 2 months of presentation (due to higher rate of nosocomial MRSA colonization)
* abcesses located on the head or neck
* children with history of a sulfa allergy
* abscesses caused by animal bite wounds
* children with Diabetes Mellitus
* abscesses arising from tattooing
* abscesses arising from vaccination sites
* pregnant females

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Resolution of abscess | 5-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pranikoff, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States